CLINICAL TRIAL: NCT06834945
Title: Addressing Fertility Information Needs and Fertility-related Distress Among Female Adult Survivors of Childhood Cancer
Brief Title: Addressing Fertility Information Needs and Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00109631; 5F32CA265054-03 (NIH)
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Childhood Cancer; Fertility Issues
Keywords: Fertility Concerns; Fertility Distress
MeSH Terms: conditions — Neoplasms; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYA SPARK (Experimental): Participants will receive the AYA SPARK health intervention which includes six sessions delivered remotely (i.e., videoconferencing) by a clinical psychologist.
  Interventions: Behavioral: AYA SPARK

INTERVENTIONS:
Behavioral: AYA SPARK — Intervention includes video conferencing based sessions to cover topics related to fertility-related information needs and concerns among female adult survivors of childhood cancer over a 6-8 week period.

SUMMARY:
The purpose of this study is to develop and refine a behavioral intervention to address fertility-related information needs and fertility-related distress among female adult survivors of childhood cancer.

DETAILED DESCRIPTION:
Adult survivors of childhood cancer are a growing population who face a number of long-term and late effects secondary to their cancer treatment, which have the potential to profoundly impact their future health, quality of life, and achievement of life goals. This project will examine the feasibility, acceptability of a novel behavioral intervention aiming to address fertility-related information needs and fertility-related distress among adult survivors of childhood cancer.

Following the Obesity-Related Behavioral Intervention Trials (ORBIT) Model of intervention development, the proposed study seeks to design and refine a behavioral intervention to address unmet fertility-related information needs and fertility-related distress among female adult survivors of childhood cancer (aged 18-44). The intervention is organized into six remotely delivered sessions integrating patient activation theory and Acceptance and Commitment Therapy (ACT) strategies, and evidence-based reproductive health information and help to empower empower survivors to make informed decisions that align with their personal values. Intervention content will be delivered to a small sample of the target population (N=30). Feasibility and acceptability, as well as examination of pre- to post-intervention patterns of change in intervention targets (primary: fertility health knowledge, fertility-related distress; secondary: psychological flexibility, patient activation, and self-efficacy), will be assessed and utilized to further refine the intervention (e.g., intervention strategies, intervention length, and delivery modality).

Although this project is focused on the late effect of impaired fertility, the intervention developed through this study has the potential to produce significant public health benefits: it could be applied to address other late effects in this population, which if left untreated, may lead to greater health complications in this growing population later in life.

ELIGIBILITY:
Inclusion Criteria:

* Currently aged 18-44
* Diagnosed with cancer at <18 years old
* Female sex
* Uncertain fertility status

Exclusion Criteria:

* Age <18
* Currently under the care of a fertility specialist
* Having a major/serious psychiatric concern (e.g., schizophrenia) as indicated by medical chart/medical provider
* Inability to provide consent.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by treatment attrition | Post-treatment, approximately 16 months
  A treatment attrition rate of ≤ 20% will be indicative of preliminary intervention feasibility.
Feasibility as measured by session attendance | Post-treatment, approximately 16 months
  A session attendance rate of ≥80% will be indicative of preliminary intervention feasibility.
Treatment acceptability as measured by Treatment Acceptability Questionnaire (TAQ) | Post-treatment, approximately 16 months
  Acceptability will be measured by the Treatment Acceptability Questionnaire (TAQ), a six-item measure assessing perceptions of an interventions acceptability, ethics, and effectiveness. Items are rated on a 7-point Likert scale, from "very unacceptable" to "very acceptable". An average score of ≥5 will be indicative of treatment acceptability.

SECONDARY OUTCOMES:
Fertility health knowledge as measured by Modified Fertility and Infertility Treatment Knowledge Score (FIT-KS) | Pre-treatment and post-treatment, approximately 16 months
  Fertility health knowledge will be assessed via modified items from the FIT-KS, a measure examining knowledge of normal reproductive function, general fertility information, treatment factors affecting fertility, infertility information, and alternative parenting options. The total score ranges from 0 to 29, where a higher score indicates greater knowledge.
Patient activation as measured by Short Form of the Patient Activation Measure | Pre-treatment and post-treatment, approximately 16 months
  The PAM is a 13-item measure used to assess survivors' knowledge, skills, and confidence that are central to managing their health and health care. Patients are asked to rate their agreement with statements about their health and health care on a 4 point scale from "strongly disagree" to "strongly agree." From these response a total PAM score is calculated on a scale of 0-100, with higher scores indicating higher levels of activation.
Self-efficacy for communicating with medical providers as measured by a modified version of the Ask, Understand, Remember Assessment (AURA) | Pre-treatment and post-treatment, approximately 16 months
  A 6-item measure assessing self-efficacy for communication in clinical encounters. Patients are asked to rate their agreement with statements related to their confidence in asking questions, understanding explanations, and remembering information on a 4 point scale from "Disagree a lot" to "agree a lot" with higher scores indicating greater confidence in patient communication abilities within a healthcare setting.
Psychological flexibility as measured by the Acceptance and Action Questionnaire-II (AAQ-II) | Pre-treatment and post-treatment, approximately 16 months
  7-item questionnaire designed to measure psychological inflexibility rated on 7-point Likert scale (1 = never true, 7 = always true); higher total scores indicate greater levels of psychological inflexibility or experiential avoidance
Fertility-related distress will be measured by the Reproductive Concerns after Cancer (RCAC)scale | Pre-treatment and post-treatment, approximately 16 months
  RCAC an 18-item scale that assesses concerns about: fertility potential, partner disclosure, child's health, personal health, acceptance, and becoming pregnant. The RCAC has been used to assess fertility-related distress among female cancer survivors. Items are rated on a five-point Likert scale ranging from 1= "Strongly disagree" to 5= "Strongly agree." with higher scores indicating greater concerns.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No